CLINICAL TRIAL: NCT07045415
Title: The Effect of Pelvic Floor Muscle Exercises on Urinary Incontinence Management and Quality of Life in Patients Undergoing Radical Prostatectomy
Brief Title: The Effect of Pelvic Floor Muscle Exercises After Radical Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Cemile Nida Kayış, Lecturer, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-41901325-200-109794
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer (Post Prostatectomy); Urinary Incontinence (UI)
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Exercise Group (Experimental): The content of the pelvic floor muscle training program has been prepared based on the guidelines of the European Association of Urology and the American Urology Association. In order to ensure that patients in the intervention group perform pelvic floor muscle exercises (PFME) correctly, verbal explanations and visual training materials will be provided in patient rooms outside of treatment hours. During the preoperative period, patients will undergo 20 minutes of one-on-one PFME training. In the postoperative period, following the removal of the urinary catheter and until discharge, patients will undergo regular daily PFME training. In addition, detailed training will be provided to patients to continue the exercise program at home for three months, and weekly telephone calls will be made to remind them of the exercises in order to support the continuity of the program.
  During discharge, patients will be given an educational brochure (brochure provided to patients at Konya City Hosp
  Interventions: Behavioral: Pelvic Floor Muscle Exercises.
- Control Group (Other): Participants will be informed about the importance of pelvic floor muscle exercises in improving quality of life, and training will be provided with the support of verbal explanations and visual educational materials.
  Interventions: Behavioral: Pelvic Floor Muscle Exercises.

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Exercises. — A structured pelvic floor muscle training (PFME) program provided by a nurse, based on EAU and AUA guidelines, consisting of 20-minute sessions delivered 3 times a week

SUMMARY:
Cancer, a major public health problem worldwide, was one of the leading causes of mortality in 2020, accounting for approximately 10 million deaths. With 1.41 million new cases reported in the same year, prostate cancer is the fourth most common cancer type globally (Ferlay et al., 2021). Prostate cancer is not only one of the most common types of cancer in men, but it also ranks second among cancer-related deaths in men worldwide (Rahnama'i et al., 2021). Radical prostatectomy (RP) is a treatment method that involves the surgical removal of the prostate gland and surrounding tissues, to stop the progression of the disease and improve the patient's quality of life (Göktas et al., 2015; Litwin and Tan, 2017). Following radical prostatectomy, a curative treatment method commonly used to prevent metastasis, mortality rates remain low; however, the procedure carries a relatively high risk of morbidity (Akarken et al., 2020; Evren and Taşcı, 2021).

The most common complication encountered by patients after RP is urinary incontinence (Choiniere et al., 2022; Rahnama'i et al., 2021). UI arises due to factors such as damage to the internal sphincter, external rhabdosphincter, and supportive structures of the urethra during surgery, as well as the involvement of the neurovascular bundle and the development of postoperative fibrosis (Castellan et al., 2023). Urinary incontinence (UI) developing after radical prostatectomy significantly reduces patients' quality of life and negatively affects their social adaptation. Therefore, understanding the factors influencing the development of UI after radical prostatectomy is of great importance in determining appropriate treatment approaches and optimizing management (Bernardes et al., 2019; Storås et al., 2020). In the literature, the incidence rates of incontinence after radical prostatectomy range from 0.8% to 87%, and these differences are attributed to various factors such as surgical technique, patient characteristics, and evaluation methods (Boorjian et al., 2012; Hodges et al., 2019; Grise et al., 2017; Pastero et al., 2017).

In the majority of patients, moderate to severe urinary incontinence is observed in the first few weeks after surgery. In some patients, this condition may persist for months or even years. Urinary incontinence can lead to various psychosocial effects such as shame, loss of self-esteem, impaired mental well-being, anxiety, relationship and sexual dysfunction, and social isolation (Kadono et al., 2016; Zachovajeviene et al., 2017). This condition has a significant impact on patients' physical, social, and emotional well-being, as well as their daily activities, and can contribute to social isolation by causing feelings of embarrassment (Castellan et al., 2023; Ouanes et al., 2022).

Nurses play an important role in the management of urinary incontinence that develops after RP. Nurses can educate patients about urinary incontinence, teach conservative treatment methods such as pelvic floor muscle exercises (PFME), and provide psychological support to make the process more manageable (Milios et al., 2019; Tosunöz et al., 2018; Wang et al., 2018). PBME is an effective method that stands out in the rehabilitation of incontinence after RP, and it is one of the most common practices aimed at increasing the strength of the pelvic floor muscles to eliminate sphincter weakness (Castellan et al., 2023; Chitre and Kulkarni, 2023; Pratiwi et al., 2020). Studies on the effectiveness of PTKE indicate that these exercises can improve patients' urinary control (Azal et al., 2022). Nurses play a significant role in promoting pelvic floor muscle health by providing information and implementing educational programs and practices to ensure that these exercises are taught and performed correctly (Jalalinia et al., 2020; Storås et al., 2020).

This study aims to evaluate the effects of preoperative and postoperative nursing interventions on urinary incontinence management and quality of life in patients who have undergone RP. In this context, the effects of nursing interventions (education, pelvic floor muscle exercises, bladder training, etc.) on urinary incontinence severity, quality of life, and patient satisfaction will be examined comparatively. The study aims to identify the most effective nursing interventions in the management of urinary incontinence after RP and to integrate these interventions into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Being 40 years of age or older Not having urinary incontinence before surgery Having undergone Radical Prostatectomy surgery due to prostate cancer Patients who did not have urinary incontinence before surgery

Exclusion Criteria:

* Patients with congenital anomalies of the urinary system, serious organ dysfunctions (liver or kidney failure, advanced heart failure, coagulopathy), neuropsychiatric disorders, presence of active infection, and history of major abdominal or pelvic surgery will not be included in the study.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary Incontinence Severity Assessed by ICIQ-SF | Baseline (preoperative), 7 days after catheter removal, 1 month, and 3 months postoperatively
  The primary outcome is the change in urinary incontinence severity following pelvic floor muscle exercises in patients undergoing radical prostatectomy. This will be measured using the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), which evaluates frequency, amount of leakage, and impact on daily life over the past 4 weeks. Scores range from 0 to 21, with higher scores indicating greater severity. This outcome was used to inform the hypothesis and sample size calculation of the study.

SECONDARY OUTCOMES:
Change in Quality of Life Assessed by King's Health Questionnaire (KHQ) | Baseline (preoperative), 7 days after catheter removal, 1 month, and 3 months postoperatively
  The secondary outcome is the change in quality of life associated with urinary incontinence, measured using the King's Health Questionnaire (KHQ). The KHQ is a validated and reliable tool assessing nine domains: general health perception, incontinence impact, role and physical limitations, social limitations, personal relationships, emotions, sleep/energy, and severity measures. Scores range from 0 to 100, with higher scores indicating poorer quality of life. This measure will complement the assessment of group differences in response to pelvic floor muscle exercise intervention.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures, including urinary incontinence scores (ICIQ-SF) and quality of life scores (KHQ), will be shared upon reasonable request. Data will be available after publication of study results and will be shared for academic and research purposes only, in compliance with ethical approvals and participant consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Indefinite (upon request)
Access Criteria: Available after study completion and upon reasonable request with no defined end date.